CLINICAL TRIAL: NCT05703217
Title: The Effects of C Mill Virtual Reality Applied Rehabilitation and Classical Rehabilitation on Gait and Balance in Parkinson's Patients: Randomized Controlled Study
Brief Title: C Mill Virtual Reality Applied Rehabilitation and Classical Rehabilitation on Gait and Balance in Parkinson's Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Romatem Bursa Hospital (Other)
Collaborators: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Nermin Çalışır, Principal İnvestigator,Head of Neurology, Romatem Bursa Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-4/1
Record Dates: First submitted 2022-10-31; First posted 2023-01-27 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease; Rehabilitation
Keywords: Parkinson Disease; Rehabilitation; Gait; Balance
MeSH Terms: conditions — Parkinson Disease | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- classical physical therapy and rehabilitation program (Active Comparator): In classical physical therapy, muscle strengthening, sitting, standing and walking exercises will be performed with physiotherapy.
  Interventions: Procedure: classical physical therapy with physiotherapy.
- virtual reality assisted walking and balance exercise program (Active Comparator): C-Mill device: It is possible to stand and walk on the treadmill. The patient is fixed to the moving band by attaching a garment made of corset-like straps, and thanks to this system, the risk of falling of the patient is prevented. There are virtual reality applications on the treadmill floor and on the giant screen opposite: ball collection It provides adaptation of walking to normal life with animal figures, forest or street images, sounds.
  Interventions: Procedure: classical physical therapy with physiotherapy.

INTERVENTIONS:
Procedure: classical physical therapy with physiotherapy. — C-Mill device: It is possible to stand and walk on the treadmill. The patient is fixed to the moving band by attaching a garment made of corset-like straps, and thanks to this system, the risk of falling of the patient is prevented. There are virtual reality applications on the treadmill floor and on the giant screen opposite: ball collection It provides adaptation of walking to normal life with animal figures, forest or street images, sounds. In classical physical therapy, muscle strengthening, sitting, standing and walking exercises will be performed with physiotherapy.
  Other Names: C mill virtual reality applied rehabilitation

SUMMARY:
In this research; the investigators would like to compare the results of patients with Parkinson's disease in the two groups who received classical physical therapy and rehabilitation program and virtual reality assisted walking and balance exercise at the beginning (1st rehabilitation day =1. day) and end of rehabilitation (21st rehabilitation day=50.day). In addition, the investigators aimed to reveal the change of gait and balance parameters by measuring the C-mill walking and balance rehabilitation device with numerical data and graphic analysis.

DETAILED DESCRIPTION:
BASIS AND JUSTIFICATION OF THE RESEARCH: : In Parkinson's patients, difficulty in walking, slowing down in movements, difficulties in starting and maintaining walking become evident in Hoehn Yahr stage 2-3-4 stages of the disease. In addition to drug therapy, physical therapy and rehabilitation applications have proven to be effective in conditions such as walking and movement restriction in Parkinson's patients. Rehabilitation with a physiotherapist, controlled home exercise programs, and robot-assisted rehabilitation practices were all found to be effective in the clinic.

EXPECTED BENEFITS AFTER THE RESEARCH: It improves the patient's daily life activities and tests of all kinds of FTR applications. With the rehabilitation the investigators will implement, the investigators will help patients to be able to walk, sit and stand up unaided and independently. The investigators expect an increase in exercise capacity, an increase in walking distance, an improvement in balance and walking, and an increase in balance and walking measurements.

RESEARCH METHOD:

1. All measurements 1st day when rehabilitation applications started and 50th day when rehabilitation applications end.
2. To evaluate whether they benefit from the applied rehabilitation; Changes in the patient's own values will be compared on the first day and the last day of rehabilitation.
3. It will be determined whether there is a difference between the scales and values between the two groups in which classical rehabilitation and C mill virtual reality applied rehabilitation.
4. In order to determine the neurological examination status of the patients:

   UPDR s-III: Unified Parkinson's Disease Rating Scale-Motor: maximum 56 points and a high score is considered bad.

   Regarding balance and walking: Tinetti test: the maximum possible score is 28, a high score is considered good.

   To measure the time it takes to get up and walk 3 meters from the seat, turn and sit in the chair that he/she started again: The time up and go test: normal value: It was determined as less than 12 seconds.

   To determine their own thoughts about the quality of life and the health of the patient: Short Form Health Survey-36: Norm values for the Turkish society have been determined, and the values received by the patients will be interpreted accordingly.

   To determine the ability to walk: Functional Ambulation Classification (FAC): A value between 0 and 5. A high score is determined as good.
5. Walking parameters:Measurements will be made with a C mill walking and balance rehabilitation device.

It is known that walking speed, walking distance, walking time, step length, and number of steps per minute decrease in Parkinson's patients. In order to measure whether there is an increase or change in these values with rehabilitation: Measurements will be made with a C mill walking and balance rehabilitation device. The following measurements will be made by walking at the speed at which the patient can walk comfortably, for a maximum of 5 minutes: Single stance phase (%), Single stance time (s), weight transfer %, right and left stride length (cm), two stride length (cm), symmetry ( %), walking distance (m), walking time (minute), walking speed (km/h), total number of steps and number of steps per minute.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:
* Women and men
* 60-80 years old Those who have been diagnosed with Parkinson's disease and are using regular drug therapy
* Hoehn Yahr Stage: 2-3-4

Hoehn-Yahr Staging:

Stage 0- No signs of disease. Stage 1- Unilateral disease. Stage 1.5- Unilateral plus axial involvement. Stage 2- Bilateral disease, no balance disorder. Stage 2.5- Mild bilateral disease recovering in the pull test. Stage 3 - Mild to moderate bilateral disease and some postural instability, physically independent.

Stage 4 - Severe disability, able to stand and walk unaided. Stage 5 - unassisted wheelchair or bed dependent. Can be mobilized without support or with minimal support

Exclusion Criteria:

Criteria for exclusion of volunteers from the study:

* psychiatric illness, dementia
* advanced vision and hearing problems
* diseases that limit walking and movement: joint disease (knee, hip joint diseases), advanced spinal stenosis, lumbar discopathy, hemiplegia
* heart failure and respiratory failure

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
UPDR s-III: Unified Parkinson's Disease Rating Scale-Motor | 1st day: when rehabilitation applications started
  In order to determine the neurological examination status of the patients: UPDR s-III: Unified Parkinson's Disease Rating Scale-Motor: maximum 56 points and a high score is considered bad
UPDR s-III: Unified Parkinson's Disease Rating Scale-Motor | 50th day: when rehabilitation applications end
  In order to determine the neurological examination status of the patients: UPDR s-III: Unified Parkinson's Disease Rating Scale-Motor: maximum 56 points and a high score is considered bad
Tinetti test | 1st day: when rehabilitation applications started
  Regarding balance and walking: Tinetti test: the maximum possible score is 28, a high score is considered good.
Tinetti test | 50th day: when rehabilitation applications end
  Regarding balance and walking: Tinetti test: the maximum possible score is 28, a high score is considered good.
The time up and go test | 1st day: when rehabilitation applications started
  To measure the time it takes to get up and walk 3 meters from the seat, turn and sit in the chair that he/she started again: The time up and go test: normal value: It was determined as less than 12 seconds.
The time up and go test | 50th day: when rehabilitation applications end
  To measure the time it takes to get up and walk 3 meters from the seat, turn and sit in the chair that he/she started again: The time up and go test: normal value: It was determined as less than 12 seconds.
Short Form Health Survey-36 | 1st day: when rehabilitation applications started
  To determine their own thoughts about the quality of life and the health of the patient: Short Form Health Survey-36: Norm values for the Turkish society have been determined, and the values received by the patients will be interpreted accordingly.
Short Form Health Survey-36 | 50th day: when rehabilitation applications end
  To determine their own thoughts about the quality of life and the health of the patient: Short Form Health Survey-36: Norm values for the Turkish society have been determined, and the values received by the patients will be interpreted accordingly.
Functional Ambulation Classification (FAC) | 1st day: when rehabilitation applications started
  To determine the ability to walk: Functional Ambulation Classification (FAC): A value between 0 and 5. A high score is determined as good.
Functional Ambulation Classification (FAC) | 50th day: when rehabilitation applications end
  To determine the ability to walk: Functional Ambulation Classification (FAC): A value between 0 and 5. A high score is determined as good.
Single stance phase (%) | 1st day: when rehabilitation applications started
  Measurements will be made with a C mill walking and balance rehabilitation device. The following measurements will be made by walking at the speed at which the patient can walk comfortably, for a maximum of 5 minutes
Single stance phase (%) | 50th day:when rehabilitation applications end
  Measurements will be made with a C mill walking and balance rehabilitation device. The following measurements will be made by walking at the speed at which the patient can walk comfortably, for a maximum of 5 minutes
single stance time (s) | 1st day: when rehabilitation applications started d
  Measurements will be made with a C mill walking and balance rehabilitation device. The following measurements will be made by walking at the speed at which the patient can walk comfortably, for a maximum of 5 minutes
single stance time (s) | 50th day: when rehabilitation applications end
  Measurements will be made with a C mill walking and balance rehabilitation device. The following measurements will be made by walking at the speed at which the patient can walk comfortably, for a maximum of 5 minutes
two stride length (cm) | 1st day: when rehabilitation applications started
  Measurements will be made with a C mill walking and balance rehabilitation device. The following measurements will be made by walking at the speed at which the patient can walk comfortably, for a maximum of 5 minutes
two stride length (cm) | 50th day :when rehabilitation applications end
  Measurements will be made with a C mill walking and balance rehabilitation device. The following measurements will be made by walking at the speed at which the patient can walk comfortably, for a maximum of 5 minutes
right stride length (cm) | 1st day: when rehabilitation applications started
  Measurements will be made with a C mill walking and balance rehabilitation device. The following measurements will be made by walking at the speed at which the patient can walk comfortably, for a maximum of 5 minutes
right stride length (cm), | 50th day: when rehabilitation applications end
  Measurements will be made with a C mill walking and balance rehabilitation device. The following measurements will be made by walking at the speed at which the patient can walk comfortably, for a maximum of 5 minutes
left stride length (cm) | 1st day: when rehabilitation applications started
  Measurements will be made with a C mill walking and balance rehabilitation device. The following measurements will be made by walking at the speed at which the patient can walk comfortably, for a maximum of 5 minutes
left stride length (cm) | 50th day: when rehabilitation applications end
  Measurements will be made with a C mill walking and balance rehabilitation device. The following measurements will be made by walking at the speed at which the patient can walk comfortably, for a maximum of 5 minutes
walking distance (m) | 1st day: when rehabilitation applications started
  Measurements will be made with a C mill walking and balance rehabilitation device. The following measurements will be made by walking at the speed at which the patient can walk comfortably, for a maximum of 5 minutes
walking distance (m) | 50th day: when rehabilitation applications end
  Measurements will be made with a C mill walking and balance rehabilitation device. The following measurements will be made by walking at the speed at which the patient can walk comfortably, for a maximum of 5 minutes
walking time (minute) | 1st day: when rehabilitation applications started
  Measurements will be made with a C mill walking and balance rehabilitation device. The following measurements will be made by walking at the speed at which the patient can walk comfortably, for a maximum of 5 minutes
walking time (minute) | 50th day: when rehabilitation applications end
  Measurements will be made with a C mill walking and balance rehabilitation device. The following measurements will be made by walking at the speed at which the patient can walk comfortably, for a maximum of 5 minutes
walking speed (km/h) | 1st day: when rehabilitation applications started
  Measurements will be made with a C mill walking and balance rehabilitation device. The following measurements will be made by walking at the speed at which the patient can walk comfortably, for a maximum of 5 minutes
walking speed (km/h) | 50th day: when rehabilitation applications end
  Measurements will be made with a C mill walking and balance rehabilitation device. The following measurements will be made by walking at the speed at which the patient can walk comfortably, for a maximum of 5 minutes
step symmetry ( %) | 1st day: when rehabilitation applications started
  Measurements will be made with a C mill walking and balance rehabilitation device. The following measurements will be made by walking at the speed at which the patient can walk comfortably, for a maximum of 5 minutes
step symmetry ( %) | 50th day: when rehabilitation applications end
  Measurements will be made with a C mill walking and balance rehabilitation device. The following measurements will be made by walking at the speed at which the patient can walk comfortably, for a maximum of 5 minutes
number of steps per minute. | 1st day: when rehabilitation applications started
  Measurements will be made with a C mill walking and balance rehabilitation device. The following measurements will be made by walking at the speed at which the patient can walk comfortably, for a maximum of 5 minutes
number of steps per minute. | 50th day: when rehabilitation applications end
  Measurements will be made with a C mill walking and balance rehabilitation device. The following measurements will be made by walking at the speed at which the patient can walk comfortably, for a maximum of 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: NERMİN ÇALIŞIR, Study Director — ROMATEM PHYSICAL THERAPY AND REHABILITATION HOSPITALS BURSA HOSPITAL; NURTEN KÜÇÜKÇAKIR, Principal Investigator — ROMATEM ROMATEM PHYSICAL THERAPY AND REHABILITATION HOSPITALS BURSA HOSPITALS BURSA HOSPITAL; SİNEM AKSELİM, Principal Investigator — BURSA CİTY HOSPİTAL PHYSICAL THERAPY AND REHABILITATION HOSPITAL; Muhammed Ali DEMİRBAĞ, Principal Investigator — ROMATEM ROMATEM PHYSICAL THERAPY AND REHABILITATION HOSPITALS BURSA HOSPITALS BURSA HOSPITAL; RAFET AKAR, Principal Investigator — ROMATEM ROMATEM PHYSICAL THERAPY AND REHABILITATION HOSPITALS BURSA HOSPITALS BURSA HOSPITAL; ŞEYDA ÖNCÜL, Principal Investigator — ROMATEM ROMATEM PHYSICAL THERAPY AND REHABILITATION HOSPITALS BURSA HOSPITALS BURSA HOSPITAL; GÖKHAN KAYA, Principal Investigator — ROMATEM ROMATEM PHYSICAL THERAPY AND REHABILITATION HOSPITALS BURSA HOSPITALS BURSA HOSPITAL; ANIL YILMAZ, Principal Investigator — ROMATEM ROMATEM PHYSICAL THERAPY AND REHABILITATION HOSPITALS BURSA HOSPITALS BURSA HOSPITAL
Locations (1):
- Romatem Romatem Physical Therapy and Rehabilitation Hospitals Bursa Hospitals Bursa Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: as a date relative to the time when summary data are published or otherwise made available (starting 7 months after publication).
Access Criteria: all the data